CLINICAL TRIAL: NCT04377243
Title: Phase II Trial of V8 in Treating Kidney Failure
Brief Title: Immunotherapy of Chronic Kidney Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Immunitor LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V8
Record Dates: First submitted 2020-05-02; First posted 2020-05-06 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Renal Failure Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: neither patients nor attending physician are aware
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- V8 850 mg (Experimental): Arm 1: Individuals with chronic kidney failure having creatinine level twice higher than normal. They will receive once daily pill of V8
  Interventions: Biological: V8
- Placebo 850 mg (Placebo Comparator): Arm: 2 Individuals with chronic kidney failure having creatinine level twice higher than normal. They will receive once daily pill of placebo
  Interventions: Biological: V8

INTERVENTIONS:
Biological: V8 — one pill per day either V8 or placebo
  Other Names: Placebo

SUMMARY:
Kidney failure can result from inflammatory renal disease in the context of autoimmunity because the kidney is targeted by host's immune response against self. There are many causes to this, but abnormal kidney function tests, i.e., BUN and creatinine, can reveal the disease. Oral delivery of kidney cells is ought to produce the immune tolerance - phenomenon is known as oral tolerance. Preliminary studies produced convincing evidence that this hypothesis holds true and has not produced any adverse side effects. Intended open label Phase II aims to confirm these findings.

ELIGIBILITY:
Inclusion Criteria:

* Baseline level of creatinine twice above normal

Exclusion Criteria:

* Baseline level of creatinine normal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-06-16 (Estimated); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Effect on creatinine | 1 month
  Change in serum creatinine level from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Immunitor LLC, Ulaanbaatar, Mongolia